CLINICAL TRIAL: NCT05182736
Title: Taking Responsible Actions in Life Evaluation
Acronym: TRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland State University (Other)
Responsible Party: Principal Investigator, Lynne Messer, Associate Professor of Public Health, Portland State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 163673
Record Dates: First submitted 2021-09-15; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy in Adolescence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Students in comparison arm received intervention as usual. Students in the comparison schools (as well as those in the intervention condition) receive the normal ninth grade health curriculum, "Reproductive and Health Safety Education," which is intended to cover three essential standards 1) Healthy and effective interpersonal communication and relationships, 2) Abstinence from sexual intercourse as a positive choice for young people, and 3) Strategies that develop and maintain reproductive and sexual health. All schools in North Carolina provide sex education in accordance with the 2009 Health Youth Act in seventh, eighth, and ninth grades
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAIL intervention (Experimental): The TRAIL program is comprised of a multi-tier system of strategies:
  1. Universal Strategies (delivered school-wide),
  2. Targeted Strategies (delivered to the target grade level in the evaluation sample)
  3. Intensive Strategies (delivered to select at-risk students)
  Interventions: Behavioral: TRAIL intervention
- Control (No Intervention): Students in the comparison schools receive the normal ninth grade health curriculum, "Reproductive and Health Safety Education."

INTERVENTIONS:
Behavioral: TRAIL intervention — The TRAIL program is comprised of a multi-tier system of strategies: Universal strategies impact the entire school via a school-wide social norms marketing campaign and school-climate change activities. School staff trainings and professional development activities focus on enhancing protective factors for students to reduce the effects of stressful life events and trauma, improving classroom management, linking students to resources, and improving the overall school climate for students and staff. Targeted strategies include an in-school curriculum and service learning component, which impact all ninth grade students at the intervention high schools and all eighth grade students at the intervention middle schools. Intensive strategies are intended for a subset of youth and their caregivers with identified increased risk-factors, and they include peer mentoring, after-school running/positive youth development programming, summer programming, and parent workshop support.
  Arms: TRAIL intervention

SUMMARY:
TRAIL is a multi-tiered school-wide intervention delivered to middle and high school aged youth. The overall goal of the TRAIL project is to decrease rates of teen births by increasing the capacity of students to make healthy decisions regarding sexual health through the use of a school-wide pregnancy prevention model. The program will be delivered to youth in eighth and ninth grade at the intervention sites.

DETAILED DESCRIPTION:
The TRAIL program is comprised of a multi-tier system of strategies:

1. Universal Strategies (delivered school-wide) Universal strategies impact the entire school via a school-wide social norms marketing campaign and school-climate change activities. A social norms marketing campaign saturates the entire high school or middle school site through monthly newsletters, posters, and video campaigns to educate students on healthy behaviors and dispel their misperceptions of peers' sexual activity. School staff trainings and professional development activities focus on enhancing protective factors for students to reduce the effects of stressful life events and trauma, improving classroom management, linking students to resources, and improving the overall school climate for students and staff. Activities include trainings to staff and teachers on trauma-informed care, positive youth development, available teen friendly resources via the Network of Care teen resource guide and app, and available support programs to the parents. Three trainings are provided to key health staff and one training is provided to the entire school staff. Healthcare linkages and referrals are measured by school nurses and reviewed by program staff to assess and address any barriers to accessing services related to teen sexual health and related healthcare services.
2. Targeted Strategies (delivered to the target grade level in the evaluation sample) Targeted strategies include an in-school curriculum and service learning component, which impact all ninth grade students at the intervention high schools and all eighth grade students at the intervention middle schools. Elevate is the in-school adolescent leadership curriculum program that provides teens with the knowledge, skills, and support they need to make healthy decisions regarding their future, including those related to sexual health. Elevate provides peer mentoring and an interactive curriculum covering topics such as setting and achieving goals; self-assessment; issues with family, friends, and self; media awareness; self-esteem; leadership; communication and negotiation skills; and future orientation. In addition, all eighth and ninth graders complete service learning projects to develop and deepen a positive attachment to the school and community. This tier includes five 90-minute sessions (7.5 hours) of classroom programing and ten hours of service learning.
3. Intensive Strategies (delivered to select at-risk students) Intensive strategies are intended for a subset of youth and their caregivers with identified increased risk-factors, and they include peer mentoring, after-school running/positive youth development programming, summer programming, and parent workshop support. Although all eighth and ninth grade students and their caregivers are eligible to receive intensive strategies, a subset identified by the schools are be targeted. Participation is always voluntary. High school and college mentors are carefully selected and trained to act as peer mentors who collaborate to raise awareness about teen health issues in the community and promote healthy decision making. These mentors assist the universal, targeted, and intensive strategy activities. TRAIL enrichment is a twenty 90-minute session comprehensive noncompetitive running program that promotes future orientation, an active lifestyle, nutritious eating, and healthy decision-making including decisions regarding sexual health for adolescents to achieve holistic health and be successful adults. Summer Advantage opportunities provide meaningful, positive, and supervised activities for youth during the summer month. Activities are made available through community partners to allow students to experience various positive youth development outlets in the community, which are related to health, education, and the arts. Parent workshops are offered to equip parents and community members with prevention education and a system to reinforce positive norms for students.

ELIGIBILITY:
Inclusion Criteria:

* Parental passive consent (parents did not withdraw consent)
* 9th grade at baseline (cohort 1) and 8th grade at baseline (cohort 2)
* English or Spanish speaking

Exclusion Criteria:

* Cognitive impairment
* Repeat students (students repeating 9th grade for cohort 1 or 8th grade for cohort 2)
* Moved out of district prior to randomization

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4261 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Participant report of having not been abstinent in the past three months at 18-month follow up assessment | At 18 month post intervention
  Reporting not having been abstinent in the past three months

IPD SHARING:
Plan to Share IPD: No